CLINICAL TRIAL: NCT06325150
Title: The Impact of Light Exposure on Cognitive Function in Classrooms
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Hanne M Hoffmann, Principal Investigator, Michigan State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00008572
Record Dates: First submitted 2024-01-17; First posted 2024-03-22 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: This study will test the effect of light emitting glasses, vs placebo, vs no-glasses to attention in college students. This is a crossover study, where participants will be randomly assigned to one of three groups, and tested in random order. The students will be tested on 2 or 3 different conditions (no glasses, placebo or light emitting glasses). The assignment to each of the groups, and the order of the intervention (+/- glasses) will be randomized.
  Note-light emitting glasses are not FDA regulated. Because light emitting glasses can change physiology, this is considered a phase 1 clinical trial.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Light glasses type 1 (Experimental): Experimental light emitting glasses.
  Interventions: Device: Light emitting glasses
- Light glasses type 2 (Placebo Comparator): Placebo light emitting glasses
  Interventions: Device: Light emitting glasses
- No glasses control (No Intervention): No glasses control group

INTERVENTIONS:
Device: Light emitting glasses — Assess the capacity of 20 min use of AYO light emitting glasses on different outcomes
  Arms: Light glasses type 1; Light glasses type 2

SUMMARY:
Humans are constantly exposed to a variety of light types, created naturally or through artificial means. Light exposure captured by the eyes impacts many physiological functions in humans, including but not limited to cognitive output, fatigue levels, and mood regulation. The level of impact on cognitive learning from different types of light on undergraduate adult students remains unclear.

DETAILED DESCRIPTION:
This study has chosen to test light's impact on adult (18 years and older) undergraduate students' cognitive function. We hypothesize that students who wear light-enriched Type1 glasses (bright light emitting glasses) for one session (20 minutes) will experience greater cognitive function, than those who either wear light-enriched Type 2 glasses(placebo light) or no glasses at all.

This study will answer the following questions:

1. After a single session (20 minutes) of wearing light-enriched glasses, on average how much did the students' cognitive function increase as compared to students without light-enriched glasses?
2. Does cognitive function increase to a comparable degree using both types of light-enriched glasses for a single session (20 minutes)?
3. Does the time of day impact the effects of light-enriched glasses during a single session (20 minutes), thus improve cognitive function?
4. Does time of day impact cognitive function for students who do not participate in light-enriched testing?

   The study will gather additional data variables on the following questions:
5. After wearing either type of light-enriched glasses, did the student's fatigue decrease throughout the study? How does this data compare to those who did not take part in light glasses testing?
6. After wearing either type of light-enriched glasses, did the student's mood increase throughout the study? How does this data compare to those who did not take part in light glasses testing?
7. How does the compiled data from the questionnaires and tests compare to sleep data collected from Smart Watches?

Objectives:

* Data points from participants will be captured through the following questionnaires and testing methods:

  1. Consent Form (~ 4 min)
  2. Student Questionnaire (~ 2 min) [Demographics]
  3. Chronotype Questionnaire, Morningness - Eveningness Self-Assessment * (~ 4 min)[This document tells you if you are an early bird or a night owl.]
  4. Pittsburgh Sleep Questionnaire* (~ 2 min) [This document tells you your sleep quality.]
  5. PHQ-9 Test * (~ 2 min) [This document assesses your mood.]
  6. PROMIS Fatigue Score Test [Measures your current fatigue levels.]
  7. Trail Making Test [Measures your cognitive function.]
* Additional data variables will be obtained from sleep data captured on personal Smart Watches by participants in the study. In the Student Questionnaire, participants are asked if they would be willing and able to provide the research team with their personal sleep data, covering a time period of two weeks prior to the study and three weeks during the study. This will enable researchers to compare Smart Watch data with fatigue scores and the Sleep Quality Index (Pittsburgh Sleep Questionnaire).
* Prior to testing, light composition readings will be taken from numerous locations within the classrooms and outdoors. Light readings will be obtained through a Spectral Light Meter. These readings will allow the researchers to control for ambient light exposure prior to the testing of the light emitting glasses.

ELIGIBILITY:
Inclusion criteria for wearing light glasses:

* Current Michigan State University (MSU) Undergraduate Student
* Are 18 years or older
* Healthy subject without light sensitivity
* Average bedtime 9:30 pm - 2:00 am, 6 out of 7 days a week
* Willingness to measure and report fatigue levels
* Willingness to participate in cognitive testing
* Willingness to wear light-enriched glasses in the classroom

Inclusion criteria for the control group (will not wear light glasses):

* Current Michigan State University (MSU) Undergraduate Student
* Are 18 years or older
* Average bedtime 9:30 pm - 2:00 am, 6 out of 7 days a week
* Willingness to measure and report fatigue levels
* Willingness to participate in cognitive testing

Inclusion criteria for the control group (will not wear light glasses):

* Current Michigan State University (MSU) Undergraduate Student
* Are 18 years or older
* Average bedtime 9:30 pm - 2:00 am, 6 out of 7 days a week
* Willingness to measure and report fatigue levels
* Willingness to participate in cognitive testing

Exclusion criteria for wearing light glasses:

* Are younger than 18 years of age
* Participation in shift work (evening/night shifts, early morning shifts, rotating shifts, etc.)
* Pregnant women
* Previous diagnosis of diabetes
* Use of medication that would cause sensitivity to light (e.g., antidepressants, antibiotics,prescribed sleep medication, prescribed pain meds)
* Epilepsy or a history of seizures
* Photophobia - sensitivity or eye discomfort to bright light
* Eye Diseases that limit the ability of light to be processed (e.g., untreated cataracts,severe glaucoma, macular degeneration, blindness, pupil dilation problems, or retinadamage)
* Previous eye surgery
* Previous head injuries (e.g., concussions)
* Current chronic, severe headaches/migraines
* Clinical insomniacs or those with diagnosed sleep disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All genders are able to participate in study.
Enrollment: 300 (Estimated)
Dates: Start 2026-05-16 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of attention | 3 weeks. One test per week
  To measure the impact of the intervention on attention, for each student we will measure the time it takes for the student to complete the provided test, and the number of errors in the test. Each student will completed the test, before and after the intervention, and the change in test score (time and errors) calculated.

SECONDARY OUTCOMES:
Determine how time of day impacts attention | 3 weeks. One test per week
  To determine how time of day impacts attention, we will reanalyze the data from "Outcome 1", and control for the time of day the students participated in the study. We will measure the time it took to complete the test, as well as the number of errors in the test.

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan State University, East Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: For 2 years after completion of project.
Access Criteria: Request directly from PI

REFERENCES:
- See also: Website of glasses used for study — https://goayo.com/?gclid=Cj0KCQiAhomtBhDgARIsABcaYyk3W1FLLK4wmxzR3VIz56o3vRqTYNdaEpYVTDKNekpufDattM9kMYEaAsVUEALw_wcB